CLINICAL TRIAL: NCT05594394
Title: Improving Charge Nurse Conflict Resolution Communication Using Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 104.NUR.2022.M
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-08

CONDITIONS: Conflict Resolution
MeSH Terms: conditions — Negotiating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Orai: Master Public Speaking — Participants will access the Orai: Master Public Speaking (Sani, Dhamani, & Gupta, 2020) platform with mobile and web-based applications. Communication skill-building moduleswill be assigned using exercises, case scenarios, and AI-assisted feedback debriefing through the Orai application.
  Participants will also complete case scenarios created with specific nursing conflict issues a charge nurse may encounter in an acute care facility. Upon completion of the competency development program, participants will complete the CMCSS to determine the effect on confidence levels and a brief survey (Appendix C) to assess the amicability of the program.

SUMMARY:
Nurses are being challenged to provide increasingly complex care with more inexperienced nurses due to higher rates of retirement and registered nurse (RN) turnover in general.

High-performing charge nurses with excellent interpersonal, conflict management, communication, and leadership competencies are vital to achieving optimal outcomes. Implementing a charge nurse leadership development program focused on improving communication competencies in conflict management situations can support a healthy work environment.

DETAILED DESCRIPTION:
Freedman (2019) asserts that "interpersonal conflict in nursing workplaces is a pervasive and complex phenomenon, with implications for patient safety and quality of care" (p.594). First-time leaders seldom receive adequate training for effective transition to leadership roles, with 60% reporting having no training (Gentry, Logan, & Tonidandel, 2014). Furthermore, many novice leaders struggle with transitioning from peer to leader, specifically related to interpersonal and communication skills (Basogul, 2020; Radovich, et al., 2011).

ELIGIBILITY:
Inclusion Criteria:

* RN Clinical Team Leader or Charge Nurse employed at MMMC

Exclusion Criteria:

* Non-employees of MMMC
* MMMC staff not in the role of Clinical Team Leader or Charge Nurse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • RN Clinical Team Leader or Charge Nurse employed at MMMC
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Charge nurses that have completed the program | September 2022 to November 2022
  The CMCSS is a validated tool, r= α=0.86, measuring nurses' confidence in managing challenging situations

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sweatt, MSN, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Mansfield Medical Center, Mansfield, Texas, United States

IPD SHARING:
Plan to Share IPD: No